CLINICAL TRIAL: NCT01779089
Title: The Safety and Efficacy of Minocycline as an Anti-Proteinuric in Diabetic Nephropathy
Brief Title: Minocycline and Proteinuria in Diabetic Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 013400
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Diabetic Nephropathy
Keywords: diabetic nephropathy; diabetic kidney disease; minocycline; proteinuria; albuminuria
MeSH Terms: conditions — Diabetic Nephropathies; cyclopia sequence; Proteinuria; Albuminuria | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental): Minocycline 100 mg po bid for 6 months
  Interventions: Drug: Minocycline 100 mg po bid for 6 months
- Placebo (Placebo Comparator): Placebo one tablet po bid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Minocycline 100 mg po bid for 6 months — Minocycline 100 mg po bid or placebo for 6 months
  Arms: Minocycline
Drug: placebo
  Arms: Placebo

SUMMARY:
Diabetic kidney disease increases the risk of illness and death from heart disease in patients with Type 2 diabetes. Some blood pressure medications called ACE inhibitors and ARBs slow progression of kidney disease, but the dose that can be used is often limited by side effects that are experienced by patients. The most limiting side effects of the current treatments are lowering of the kidney function or blood pressure, and a rise in blood potassium levels. A safe and inexpensive medication that doesn't lower kidney function or blood pressure or raise serum potassium would be useful.

Minocycline is a tetracycline antibiotic with recently appreciated protective properties. In a published journal article by Dr. Isermann, minocycline prevented the death of specialized kidney cells in mice. The kidneys of these mice did not develop diabetic kidney disease when seen under the microscope and the mice experienced only a little bit of protein loss in the urine. In a different published paper, the authors showed that minocycline also decreased kidney injury in a model of non-diabetic kidney disease. A related tetracycline antibiotic was shown to lower urine protein in diabetic patients. These data support a rationale for testing to see if minocycline is safe and helpful in patients with diabetic kidney disease. In this study, all patients will stay on their usual medications for the treatment of diabetic kidney disease. Patients will be given either minocycline (100 mg by mouth twice a day for 24 weeks) or placebo (an inactive capsule taken twice a day for 24 weeks). Minocycline or placebo will be assigned by a process called "randomization", which is like a coin toss. Neither the patient nor the study team will know if the patient is taking placebo or minocycline until the end of the study. The study will assess minocycline safety and test to see if minocycline is helpful or not helpful for the treatment of diabetic kidney disease.

This study was funded by the American Diabetes Association and is not supported by any pharmaceutical company.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes and diabetic nephropathy as described in the Family Investigation of Nephropathy and Diabetes Protocol
* Baseline creatinine clearance > 30 mL/min/1.73 m2 (at first screening visit)
* Proteinuria ≥ 1.0 g/day (at first screening visit)
* Age ≥30 years
* BP at baseline <150/95 mm Hg (measured sitting after 10 min rest at first screening visit)
* Adequate hepatic function defined as total bilirubin < 1.5 x the upper limit of the normal range (ULN), AST (SGOT) and ALT (SGPT) < 2.5 x ULN.
* Patients taking ACEi, angiotensin receptor blockers (ARBs), aliskerin, spironolactone and/or diltiazem may be entered, but dosing may not change during the period of study or within 1 month prior to the first of the baseline proteinuria measurements.

Exclusion Criteria:• NSAID (including COX-2 inhibitors) use > 3 tabs/week habitually

* Diagnosis of neurodegenerative diseases (Parkinson's disease, Huntington's disease, multiple sclerosis, Alzheimer's disease, etc).
* Any unstable medical illness (unstable angina, advanced cancer, etc) over the last 30 days.
* History of liver disease (screening AST > 3 times the upper limit of normal)
* History of hematologic disease (screening white blood cell count less than 3,800/mm3)
* History of systemic vasculitis or systemic lupus erythematosus
* Treatment with procainamide or hydralazine
* History of vestibular disease (excluding benign position vertigo)
* Pregnancy or lactation
* Allergy to tetracycline antibiotics
* Use of minocycline within thirty days of baseline visit
* Use of anti-epileptic medications other than gabapentin
* Use of lithium, digoxin, warfarin, other anticoagulants, and theophylline
* Limited mental capacity rendering the subject unable to provide written informed consent or comply with evaluation procedures
* History of recent alcohol or drug abuse or noncompliance with treatment or other experimental protocols
* Use of any investigational drug within 30 days prior to the baseline visit
* Women with the potential to become pregnant who are not willing to practice double-barrier birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in 24 hour urine protein/creatinine ratio (average of 2 values) baseline compared to 6-months in placebo vs minocycline | 6 months

SECONDARY OUTCOMES:
Change in average MACR in 24 hour urine, daytime and overnight collections (baseline vs 6 mos) | 6 months
Change in average 24 hour urine protein/creatinine in daytime vs overnight collections, baseline vs 6 mos | 6 mos
Change in urine and blood biomarkers in minocycline vs placebo treated patients at baseline vs 6 mos | 6 mos

OTHER OUTCOMES:
Safety | 6 mos
  Track the development of positive ANA and ANCA in placebo and minocycline-treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Sharon G Adler, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Reaearch Institute at Harbor-UCLA Medical Center, Torrance, California, United States

REFERENCES:
- [Derived] Shah AP, Shen JI, Wang Y, Tong L, Pak Y, Andalibi A, LaPage JA, Adler SG. Effects of Minocycline on Urine Albumin, Interleukin-6, and Osteoprotegerin in Patients with Diabetic Nephropathy: A Randomized Controlled Pilot Trial. PLoS One. 2016 Mar 28;11(3):e0152357. doi: 10.1371/journal.pone.0152357. eCollection 2016. PMID 27019421